CLINICAL TRIAL: NCT05031585
Title: A Pivotal, Double-blind, Parallel, Randomized, Multicenter, Superiority Clinical Trial to Evaluate the Efficacy and Safety of Nasal Lubricant Compared to Placebo on Snoring
Brief Title: Efficacy and Safety Study of Nasal Lubricant Compared to Placebo on Snoring
Acronym: RONCO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brainfarma Industria Química e Farmacêutica S/A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HYP 002-21
Record Dates: First submitted 2021-08-10; First posted 2021-09-02 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-03

CONDITIONS: Snoring; Sleep Disorder
Keywords: nasal lubricant; sleep; medical device
MeSH Terms: conditions — Snoring; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Nasal lubricant spray
  Interventions: Device: Roncoliv
- Placebo (Placebo Comparator): Placebo spray
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Roncoliv — The medical device with nasal spray solution should be used 1 time a day, before bedtime, for 30 days.
  Arms: Intervention Group
Device: Placebo — The medical device with placebo should be used 1 time a day, before bedtime, for 30 days.
  Arms: Placebo

SUMMARY:
Pivotal clinical trial, multicenter of superiority, randomized, double-blind, parallel groups, placebo-controlled and use of nasal lubricant on snoring.

DETAILED DESCRIPTION:
This study is designed for the improvement of snoring, characterized by a noise caused by the vibration of tissues obstructing the nasopharynx and oropharynx during sleep.

It is performed in participants of both sexes, over 18 years of age, who complain of snoring.

The rationale for studying the use of a medical device with nasal spray solution for snoring improvement is due to the fact that surface tension in the pharyngeal mucosa plays an important role in determining airway collapsibility.

ELIGIBILITY:
Inclusion Criteria:

* Have signed the informed consent form;
* Participants of both genders aged ≥ 18 years;
* Report of snoring assessed objectively through the standardized criteria in the snoring noise domain in the Berlin questionnaire;

Exclusion Criteria:

* History of allergy or hypersensitivity to the components of the nasal lubricant;
* Fixed nasal obstruction;
* Upper Airway Infections active or present for less than 7 days;
* Use of benzodiazepines and sleep inducing drugs;
* Under treatment for sleep apnea of any modality currently or within the past 6 months;
* Hepatic insufficiency;
* Active neoplastic disease;
* Severe sleep apnea determined by polysomnography (AHI > 30);
* Moderate sleep apnea with presence of excessive daytime sleepiness;
* Clinically significant illness or surgery, at the discretion of the principal investigator, within 30 days prior to study inclusion;
* History of chemical dependence or alcohol abuse;
* Any neurological and psychiatric disease or significant laboratory finding present, unless adequately controlled with medication allowed in the protocol;
* Patients with laboratory tests of SGOT, SGTP or CPK increased by at least two times the upper value of normal at the time of study inclusion;
* Women who are pregnant or breastfeeding or who have the desire to become pregnant;
* History of infarction and stroke;
* Craniofacial malformation;
* BMI > 35 Kg/m2;
* IDO ≥ 30 events/h determined in residence by Biologix®;
* Have symptoms of COVID-19 (fever, cold, loss of smell, loss of taste, dry cough, sore throat, diarrhea, difficulty breathing, fatigue, body aches and pains, headache).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
The effect of nasal lubricant in the improvement of snoring when compared to placebo. | 30 days of medical device use
  For the primary endpoint, the level of continuous noise equivalent to the sound produced during sleep - LAeqT (equivalent-continuous sound pressure level), in dB(A), with a frequency filter in the weighting (sound level meter - Fusion SLM®) will be evaluated.

SECONDARY OUTCOMES:
The effect of nasal lubricant on snoring reduction during polysomnography | 30 days of medical device use
  Qualitative noise evaluation through standardized algorithm with maximum noise peak (in dB), evaluated by Fusion SLM® sound level meter; Evaluation of oximetry, through Biologix®
Nasal lubricant on snoring reduction during polysomnography | 30 days of medical device use
  Quantitative noise evaluation through standardized algorithm with maximum noise peak (in dB), evaluated by Fusion SLM® sound level meter; Evaluation of oximetry, through Biologix®
Perception of snoring reduction by the partner | 30 days of medical device use
  Questioning during medical consultation
The effect of nasal lubricant on apnea observed on polysomnography | 30 days of medical device use
  Apnea and hypopnea index
The effect of nasal lubricant on sleep quality using the standardized daytime sleepiness assessment questionnaire | 30 days of medical device use
  Epworth Sleepiness Scale (ESS) measures the chance of dozing on a scale of 0 to 3, 0 being no chance and 3 being a great chance.
The effect of nasal lubricant on sleep quality using the standardized Sleep Apnea Quality Life Index (SAQLI) questionnaire | 30 days of medical device use
The effect of nasal lubricant on sleep quality using the Berlin Questionnaire / STOP-BANG Questionnaire | 30 days of medical device use
The effect of nasal lubricant on oximetry, in residence using Biologix®. | Through study completion, an average of 30 days
The effect of nasal lubricant on snoring index, in residence using Biologix®. | Through study completion, an average of 30 days

OTHER OUTCOMES:
Adverse event rate, evaluated from questioning or spontaneous reporting of serious and non-severe adverse events and findings on clinical examinations. | Through study completion, an average of 30 days
General participant well-being. | Through study completion, an average of 30 days
  Questioning during medical consultation

CONTACTS AND LOCATIONS:
Overall Officials: Brainfarma Indústria Química Farmacêutica, Study Director — Brainfarma Industria Química e Farmacêutica S/A
Locations (1):
- Núcleo Interdisciplinar Da Ciencia Do Sono, São Paulo, Brazil